CLINICAL TRIAL: NCT05353634
Title: Research on the Diagnostic Application of Metagenomic Sequencing in Clinical Infectious Diseases
Brief Title: Metagenomic Sequencing in Clinical Infectious Diseases
Status: Completed | Type: Observational
Sponsor: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022097
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Bacterial Infections and Mycoses
Keywords: clinical metagenomics; infection diseases
MeSH Terms: conditions — Bacterial Infections and Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected patients with mNGS: If the patient is suspected of infection, mNGS is performed for testing.
  Interventions: Diagnostic Test: Effects of mNGS on infected patients
- Infected patients without mNGS: The patient is suspected of being infected, and no mNGS test was performed, only other tests were performed.
  Interventions: Diagnostic Test: Effects of mNGS on infected patients

INTERVENTIONS:
Diagnostic Test: Effects of mNGS on infected patients — The impact of mNGS on infected patients, including diagnostic value, drug selection, treatment prognosis, economic burden, etc.

SUMMARY:
Progress in the diagnosis of infectious pathogens depends on the development of effective methods and the discovery of suitable biomarkers. There are several kinds of methods that have been used in diagnosis of various pathogens, such as microscopic examination, culture, serologic diagnosis or molecular approaches, etc. However, these methods have similar limitations, that is, the single detection of reagents. More importantly, physicians seldom consider infections with rare pathogens. Recently developed metagenomic next-generation sequencing (mNGS) has the capability to overcome limitations of traditional diagnostic tests. This new technology could identify all pathogens directly from sample with a single run in a hypothesis-free and culture-independent manner. Studies have shown that mNGS is more sensitive than traditional culture method in clinical conditions such as blood stream, respiratory and general infections. More importantly, due to unbiased sampling, mNGS is theoretically able to identify not only known but also unexpected pathogens or even discovery novel organisms. It should be noted that mNGS also has some limitations such as human genome contamination and possibly environmental microbial contamination. The vast majority of reads in mNGS are derived from human host. This would impede the overall analytical sensitivity of mNGS for pathogen detection. Host depletion methods or targeted sequencing may help to partially mitigate this disadvantage. As mNGS could not, by itself, define whether the detected microbe is the causative pathogen or environmental microorganism, a multidisciplinary discussion by clinicians, microbiologists as well as the lab technicians is required to interpret the result.

ELIGIBILITY:
Inclusion Criteria:

* All the patients have received mNGS testing in clinical practice.

Exclusion Criteria:

* Interruption of patient treatment process and incomplete information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the enrolled patients have received mNGS testing in clinical practice. Clinical data were rigorously evaluated and summarized, patients' data were compiled until death or hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 2022097 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Receiver operating characteristic (ROC) curves evaluate the performance of mNGS and traditional microbiological testing | From admission to discharge, 3 weeks
  Receiver operating characteristic (ROC) curves were used to evaluate the performance of the logarithm of reads per kilobase per million mapped reads [lg(RPKM)], genomic coverage, and relative abundance of the organism in predicting the true-positive pathogenic bacteria. Clinical data were rigorously evaluated and summarized to identify promising clinical indices and limitations of the mNGS-based test.

CONTACTS AND LOCATIONS:
Overall Officials: Shengjun Ma, Dr., Study Chair — Liaocheng People's Hospital
Locations (1):
- Liaocheng People's Hospital, Liaocheng, Shandong, China

IPD SHARING:
Plan to Share IPD: No